CLINICAL TRIAL: NCT03763656
Title: A Prospective Open Label, Pharmacokinetic Study of an Oral Hydroxyurea Solution in Children With Sickle Cell Anemia.
Brief Title: Pharmacokinetics of Oral Hydroxyurea Solution
Acronym: HUPK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INV543; 2017-004568-37 (EudraCT Number)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Sickle Cell Disease; Sickle-Cell; Hemoglobin Disease, Thalassemia; Sickle Cell-beta-thalassemia; Sickle Cell Hemoglobin C
Keywords: Hydroxyurea; Hydroxycarbamide; Xromi
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; Thalassemia; Hemoglobin SC Disease | interventions — Hydroxyurea; Solutions

STUDY DESIGN:
Intervention Model Description: Open label, observational, pharmacokinetic study of oral hydroxyurea solution administered to children from 6 months-17.99 years over a 12-15-month period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Novel oral solution formulation of hydroxyurea
  Interventions: Drug: Oral Hydroxyurea (100 mg/mL) Solution

INTERVENTIONS:
Drug: Oral Hydroxyurea (100 mg/mL) Solution — Participants received Oral Hydroxyurea 15 mg/kg once daily. Escalated by 5 mg/kg/day every 8-12 weeks until maximum tolerated dose achieved, up to a maximum 35 mg/kg/day.

SUMMARY:
An open label, safety and pharmacokinetic study of oral hydroxyurea solution administered to children from 6 months to 17.99 years (i.e. to the day before 18th birthday), with a 12 to 15 month treatment period for each participant. The study treatment duration will be for 6 months at the maximum tolerated dose [MTD], which is usually reached by 6 months after initiation of treatment. For patients in whom time to MTD is longer than 6 months or not achieved at all, the maximum duration of study treatment will be 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged from 6 months to 17.99 years of age (i.e. to the day before 18th birthday).
2. Diagnosis of sickle cell anemia (HbSS and HbSβº).
3. Parent(s)/legal guardian able and willing to provide written informed consent for the child to take part in the study.
4. Where applicable, the child should assent to undergo blood sampling for pharmacokinetic and biochemistry purposes and to allow physiological measurements to be made.

Exclusion Criteria:

1. Any clinically significant medical condition or abnormality, which, in the opinion of the Investigator, might have compromised the safety of the patient or which might have interfered with the study.
2. Hydroxyurea use within 6 months before enrolment.
3. Renal insufficiency (known creatinine more than twice the upper limit of normal (ULN) for age and >1.0 mg/dL [88.4 μmol/L]).
4. Clinical evidence of hepatic compromise with alanine aminotransferase (ALT) >3 times the ULN (a temporary swing in ALT did not result in exclusion).
5. Other significant organ system dysfunction based on the site Investigators discretion.
6. Severe active infections: fungal, viral or bacterial (as confirmed by culture), examples included tuberculosis, malaria, active hepatitis, osteomyelitis or any other illness that would have precluded the use of HU in normal clinical practice.
7. Active chronic leg ulcers.
8. Known allergy to oral HU solution or any of the excipients.
9. Positive pregnancy test for females of child-bearing potential (in post-menarcheal females) before initiation of treatment, unless participant was sexually abstinent. Note: True abstinence was considered as being in line with the preferred and usual lifestyle of the participant. Periodic abstinence (such as calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
10. Inadequate contraception measures in sexually active females (post-menarcheal females) and males of child-bearing age (see Section 9.5.1.10.4).
11. Breastfeeding at study initiation.
12. Participation in another clinical trial of an IMP.
13. Known infection with HIV.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela E Rankine- Mullings, MD, Principal Investigator — University of the West Indies, Mona, Kingston, Jamaica
Locations (6):
- Dr Angela E Rankine- Mullings, Kingston, Jamaica
- United Kingdom (5):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Evelina London Children's Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - The Royal London Children's Hospital, Barts Health NHS Trust, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one Jamaican sickle cell clinic (n=12) and five UK hospitals (n=20). The first participant was enrolled on 03 Jan 2019 and the last participant was enrolled on 16 Dec 2020.
Pre-assignment Details: 33 participants enrolled met the inclusion criteria; 32 initiated treatment with open label Hydroxyurea and one participant discontinued pre-treatment.
Groups:
- Oral Hydroxyurea: Participants received Oral Hydroxyurea 15 mg/kg once daily. Escalated by 5 mg/kg/day every 8-12 weeks until maximum tolerated dose achieved, up to a maximum 35 mg/kg/day.
  Hydroxyurea: Oral Hydroxyurea 100 mg/ml solution
Period: Overall Study
Arm/Group | Oral Hydroxyurea
Started (Overall (Screened)) | 33 (36 Participants were screened but 33 enrolled)
Pre-treatment Discontinuation | 1 (1 participant discontinued prior to treatment initiation. The participant was excluded from the safety population but was included in some baseline data.)
Safety Population | 32 (32 participants (split into age categories of 6months-1.99 years, 2-5.99 years and 6-17.99 years) were included in the safety population and initiated treatment with hydroxyurea.)
Age Group (6 Months - 1.99 Years) | 6
Discontinuations From Age Group (6 Months - 1.99 Years) | 3 (Reasons for discontinuation: n=1 physician decision n=2 other (participants decision not to continue))
Completed From Age Group (6 Months - 1.99 Years) | 3
Age Group (2 - 5.99 Years) | 16
Discontinuations From Age Group (2 - 5.99 Years) | 2 (Reason for discontinuation: n=2 other (migrated; participants decision to withdraw unwilling to travel))
Completions From Age Group (2 - 5.99 Years) | 14
Age Group (6 - 17.99 Years) | 10
Discontinuations From Age Group (6 - 17.99 Years) | 3 (Reason for discontinuation: n=1 protocol deviation n=2 other (participant unwilling to continue, non compliant))
Completions From Age Group (6 - 17.99 Years) | 7
Completed (Overall from all age groups) | 24
Not Completed | 9
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Participant demographics were summarized for all 33 participants. One participant discontinued prior to receiving a first dose of IMP. The remaining safety population consisted of 32 participants who all received at least one dose of the IMP and one valid primary efficacy PK measurement. This safety population was used for all analyses of baseline characteristics, secondary and exploratory outcomes, as well as safety outcomes.
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 33
Age, Customized [Count of Participants; unit: Participants]
  Age by Category: Age Group (6 months - 1.99 years) | 6
  Age by Category: Age Group (2 - 5.99 years) | 16
  Age by Category: Age Group (6 - 17.99 years) | 11
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Overall demographic population of 33 participants.
  Participants
    Sex: Female, Male (Overall): Female | 17
    Sex: Female, Male (Overall): Male | 16
    Sex: Female, Male (Age group 6 months - 1.99 years): number analyzed (Participants) | 6
    Sex: Female, Male (Age group 6 months - 1.99 years): Female | 5
    Sex: Female, Male (Age group 6 months - 1.99 years): Male | 1
    Sex: Female, Male (Age group 2 - 5.99 years): number analyzed (Participants) | 16
    Sex: Female, Male (Age group 2 - 5.99 years): Female | 5
    Sex: Female, Male (Age group 2 - 5.99 years): Male | 11
    Sex: Female, Male (Age group 6 - 17.99 years): number analyzed (Participants) | 11
    Sex: Female, Male (Age group 6 - 17.99 years): Female | 7
    Sex: Female, Male (Age group 6 - 17.99 years): Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall demographic population of 33 participants.
  Participants
    Ethnicity Overall: Hispanic or Latino | 0
    Ethnicity Overall: Not Hispanic or Latino | 33
    Ethnicity Overall: Unknown or Not Reported | 0
    Ethnicity (Age Group 6 months - 1.99 years): number analyzed (Participants) | 6
    Ethnicity (Age Group 6 months - 1.99 years): Hispanic or Latino | 0
    Ethnicity (Age Group 6 months - 1.99 years): Not Hispanic or Latino | 6
    Ethnicity (Age Group 6 months - 1.99 years): Unknown or Not Reported | 0
    Ethnicity (Age Group 2 - 5.99 years): number analyzed (Participants) | 16
    Ethnicity (Age Group 2 - 5.99 years): Hispanic or Latino | 0
    Ethnicity (Age Group 2 - 5.99 years): Not Hispanic or Latino | 16
    Ethnicity (Age Group 2 - 5.99 years): Unknown or Not Reported | 0
    Ethnicity (Age Group 6 - 17.99 years): number analyzed (Participants) | 11
    Ethnicity (Age Group 6 - 17.99 years): Hispanic or Latino | 0
    Ethnicity (Age Group 6 - 17.99 years): Not Hispanic or Latino | 11
    Ethnicity (Age Group 6 - 17.99 years): Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Overall demographic population of 33 participants. This has been further subdivided to give the demographic per age group.
  All participants identified as Black or African American except for two UK participants who self-described as Other: "Caribbean" [sic] and "Black British".
  Participants
    Race (Overall): American Indian or Alaska Native | 0
    Race (Overall): Asian | 0
    Race (Overall): Black or African American | 31
    Race (Overall): Native Hawaiian or Other Pacific Islander | 0
    Race (Overall): White | 0
    Race (Overall): Other (Specify): [sic] Caribbean | 1
    Race (Overall): Other (Specify): Black British | 1
    Race (Age Group 6 months - 1.99 years): number analyzed (Participants) | 6
    Race (Age Group 6 months - 1.99 years): American Indian or Alaska Native | 0
    Race (Age Group 6 months - 1.99 years): Asian | 0
    Race (Age Group 6 months - 1.99 years): Black or African American | 5
    Race (Age Group 6 months - 1.99 years): Native Hawaiian or Other Pacific Islander | 0
    Race (Age Group 6 months - 1.99 years): White | 0
    Race (Age Group 6 months - 1.99 years): Other (Specify): [sic] Caribbean | 1
    Race (Age Group 6 months - 1.99 years): Other (Specify): Black British | 0
    Race (Age Group 2 - 5.99 years): number analyzed (Participants) | 16
    Race (Age Group 2 - 5.99 years): American Indian or Alaska Native | 0
    Race (Age Group 2 - 5.99 years): Asian | 0
    Race (Age Group 2 - 5.99 years): Black or African American | 15
    Race (Age Group 2 - 5.99 years): Native Hawaiian or Other Pacific Islander | 0
    Race (Age Group 2 - 5.99 years): White | 0
    Race (Age Group 2 - 5.99 years): Other (Specify): [sic] Caribbean | 0
    Race (Age Group 2 - 5.99 years): Other (Specify): Black British | 1
    Race (Age Group 6 - 17.99 years): number analyzed (Participants) | 11
    Race (Age Group 6 - 17.99 years): American Indian or Alaska Native | 0
    Race (Age Group 6 - 17.99 years): Asian | 0
    Race (Age Group 6 - 17.99 years): Black or African American | 11
    Race (Age Group 6 - 17.99 years): Native Hawaiian or Other Pacific Islander | 0
    Race (Age Group 6 - 17.99 years): White | 0
    Race (Age Group 6 - 17.99 years): Other (Specify): [sic] Caribbean | 0
    Race (Age Group 6 - 17.99 years): Other (Specify): Black British | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20
  Jamaica | 13
SCA Type [Count of Participants; unit: Participants] — Measure Analysis Population Description: SCD Genotype of overall demographic population of 33 participants. Population: SCD Genotype of overall demographic population of 33 participants. SCD is caused by a mutation in the β-globin gene HBB. Hemoglobin SS (HbSS) represents a large proportion of SCD in the Americas, UK, and certain regions of Africa while higher proportions of hemoglobin SC are observed in Burkina Faso and hemoglobin Sβ-thalassemia (HbS/β0 or HbS/β+) in Greece and India. Patients with HbSS and HbS/βo-thalassaemia typically have a more severe course of disease than other genotypes.
  Participants
    SCA Type (Overall): HbSS | 32
    SCA Type (Overall): HbSbeta0 | 1
    SCA Type (Age Group 6 months - 1.99 years): number analyzed (Participants) | 6
    SCA Type (Age Group 6 months - 1.99 years): HbSS | 6
    SCA Type (Age Group 6 months - 1.99 years): HbSbeta0 | 0
    SCA Type (Age Group 2 - 5.99 years): number analyzed (Participants) | 16
    SCA Type (Age Group 2 - 5.99 years): HbSS | 15
    SCA Type (Age Group 2 - 5.99 years): HbSbeta0 | 1
    SCA Type (Age Group 6 - 17.99 years): number analyzed (Participants) | 11
    SCA Type (Age Group 6 - 17.99 years): HbSS | 11
    SCA Type (Age Group 6 - 17.99 years): HbSbeta0 | 0
Height [Mean (Standard Deviation); unit: cm] — Height in (cm) for safety population at baseline, defined as the last non-missing measurement prior to first exposure to oral hydroxurea. Population: Overall safety population of 32 participants, data available at screening for 31 participants.
  Height or length was unobtainable for 1 participant who was under the age of 2 years (Age group 6 months - 1.99 years).
  cm
    Height (cm) (Overall): number analyzed (Participants) | 31
    Height (cm) (Overall) | 109.26 (26.038)
    Height (cm) Age Group (6 months - 1.99 years): number analyzed (Participants) | 5
    Height (cm) Age Group (6 months - 1.99 years) | 79.40 (5.237)
    Height (cm) Age Group (2 - 5.99 years): number analyzed (Participants) | 16
    Height (cm) Age Group (2 - 5.99 years) | 98.08 (6.947)
    Height (cm) Age Group (6 - 17.99 years): number analyzed (Participants) | 10
    Height (cm) Age Group (6 - 17.99 years) | 142.09 (15.872)
Weight [Mean (Standard Deviation); unit: kg] — Weight in (kg) for safety population at baseline, defined as the last non-missing measurement prior to first exposure to oral hydroxyurea. Population: Overall safety population of 32 participants.
  kg
    Weight (kg) Overall: number analyzed (Participants) | 32
    Weight (kg) Overall | 19.63 (10.955)
    Weight (kg) Age Group (6 months - 1.99 years): number analyzed (Participants) | 6
    Weight (kg) Age Group (6 months - 1.99 years) | 11.18 (1.017)
    Weight (kg) Age Group (2 - 5.99 years): number analyzed (Participants) | 16
    Weight (kg) Age Group (2 - 5.99 years) | 14.74 (2.092)
    Weight (kg) Age Group (6 - 17.99 years): number analyzed (Participants) | 10
    Weight (kg) Age Group (6 - 17.99 years) | 32.52 (11.441)

OUTCOME MEASURES:

1. Primary Outcome: Clearance (CL/F)
Description: Model estimated Pharmacokinetic Parameter (PK population: n=32, having received at least one dose of study drug).
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 12 hours post-dose on Day 1 and Day 2 (Week 20-36)
Population: Clearance value for patient of 15.05 kg
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
L/hr | 3.61 [3.29 to 3.92]

2. Primary Outcome: Volume of Distribution (V/F)
Description: Model estimated Pharmacokinetic Parameter (PK population: n=32, having received at least one dose of study drug).
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 12 hours post-dose on Day 1 and Day 2 (Week 20-36)
Population: Volume of distribution for central and peripheral compartments for patient of 15.05 kg
Measure: Mean (95% Confidence Interval); unit: L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
L | 11.4 [9.52 to 13.2]

3. Primary Outcome: Time to Maximum Concentration (Tmax)
Description: Mean Tmax (h) pharmacokinetic parameter derived using the final population PK model.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 12 hours post-dose on Day 1 and Day 2 (Week 20-36)
Population: PK population = 32 participants, who have received at least one dose at 15 mg/kg and have at least one sample of PK plasma above the lower limit of quantification
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
hours
  Tmax (Overall) | 1.253 (0.412)
  Tmax (Age Group 6 months - 1.99 years): number analyzed (Participants) | 6
  Tmax (Age Group 6 months - 1.99 years) | 1.265 (0.322)
  Tmax (Age Group 2 - 5.99 years): number analyzed (Participants) | 16
  Tmax (Age Group 2 - 5.99 years) | 1.238 (0.455)
  Tmax (Age Group 6 - 17.99 years): number analyzed (Participants) | 10
  Tmax (Age Group 6 - 17.99 years) | 1.269 (0.423)

4. Primary Outcome: Maximum Plasma Concentration Cmax (ug/mL)
Description: Mean Cmax (ug/mL) pharmacokinetic parameter derived using the final population PK model.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 12 hours post-dose on Day 1 and Day 2 (Week 20-36)
Population: PK population: n=32 safety population, having received at least one dose of study drug at 15mg/kg and one sample of PK plasma above the lower limit of quantification.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
ug/mL
  Cmax (Overall) | 13.124 (1.742)
  Cmax (Age Group 6 months - 1.99 years): number analyzed (Participants) | 6
  Cmax (Age Group 6 months - 1.99 years) | 12.807 (1.399)
  Cmax (Age Group 2 - 5.99 years): number analyzed (Participants) | 16
  Cmax (Age Group 2 - 5.99 years) | 13.068 (1.939)
  Cmax (Age Group 6 - 17.99 years): number analyzed (Participants) | 10
  Cmax (Age Group 6 - 17.99 years) | 13.404 (1.714)

5. Primary Outcome: Area Under Plasma Concentration Time Curve (AUC 0-Inf)
Description: Mean AUC 0-Infinity (hr*ug/mL) pharmacokinetic parameters derived using the final population PK model.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 12 hours post-dose on Day 1 and Day 2 (Week 20-36)
Population: PK population = 32 participants receiving at least one dose of 15mg/kg hydroxyurea and have at least one PK plasma sample above lower limit of quantification.
Measure: Mean (Standard Deviation); unit: hr*ug/mL
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
hr*ug/mL
  AUC Infinity (Overall) | 64.721 (9.339)
  AUC Infinity (Age Group 6 months - 1.99 years): number analyzed (Participants) | 6
  AUC Infinity (Age Group 6 months - 1.99 years) | 62.537 (9.016)
  AUC Infinity (Age Group 2 - 5.99 years): number analyzed (Participants) | 16
  AUC Infinity (Age Group 2 - 5.99 years) | 62.899 (7.373)
  AUC Infinity (Age Group 6 - 17.99 years): number analyzed (Participants) | 10
  AUC Infinity (Age Group 6 - 17.99 years) | 68.948 (11.649)

6. Primary Outcome: Terminal Half-life (Hours)
Description: Mean Terminal Half-life (hours) pharmacokinetic parameter derived using the final population PK model.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 12 hours post-dose on Day 1 and Day 2 (Week 20-36)
Population: PK Population n=32 where all subjects received at least one dose of 15 mg/kg hydroxyurea and have at least one sample of PK plasma above the lower limit of quantification.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
hours
  Terminal Half-life (Overall) | 3.880 (0.3004)
  Terminal Half-life (Age Group 6 months - 1.99 years): number analyzed (Participants) | 6
  Terminal Half-life (Age Group 6 months - 1.99 years) | 4.107 (0.187)
  Terminal Half-life (Age Group 2 - 5.99 years): number analyzed (Participants) | 16
  Terminal Half-life (Age Group 2 - 5.99 years) | 3.949 (0.257)
  Terminal Half-life (Age 6 - 17.99 years): number analyzed (Participants) | 10
  Terminal Half-life (Age 6 - 17.99 years) | 3.634 (0.268)

7. Secondary Outcome: Adverse Events
Description: Incidence of Adverse events during the course of the trial from screening to final follow up phone call at Week 64.
  Relatedness refers to 'at least possibly related to the IMP', with severity/toxicity assessed using the CTCAE Toxicity Grade and seriousness based on the standard definition for SAE in accordance with GCP. With the exception of SCA related events, requiring >7day hospitalisation, or extension of hospitalisation before being reported as an SAE due to their frequency within the disease population. All other non-SCA related SAEs were reportable.
Time Frame: Screening Up to Week 64
Population: Safety population n=32. Overall 339 AEs in 31 participants recorded. 7 adverse events included in this list of 339 were defined as 'Serious' as per the protocol definition (i.e. SCA related and >7days hospitalisation). A separate SAE report was made at that time with a clearly defined start and end date to be able to denote a resolution to the 'seriousness' criteria as this is an ongoing chronic condition.
Measure: Number; unit: events
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
events
  Any Adverse Events (Overall): number analyzed (Participants) | 31
  Any Adverse Events (Overall) | 339
  Treatment Emergent Adverse Events (TEAEs) Overall: number analyzed (Participants) | 31
  Treatment Emergent Adverse Events (TEAEs) Overall | 339
  Serious AEs: number analyzed (Participants) | 6
  Serious AEs | 7
  Grade >or=3 TEAEs: number analyzed (Participants) | 12
  Grade >or=3 TEAEs | 19
  Related TEAEs: number analyzed (Participants) | 9
  Related TEAEs | 28
  Commonly occurring unrelated TEAE: SCA with Crisis: number analyzed (Participants) | 18
  Commonly occurring unrelated TEAE: SCA with Crisis | 53
  Commonly occurring unrelated TEAE: Upper Respiratory Tract Infection: number analyzed (Participants) | 17
  Commonly occurring unrelated TEAE: Upper Respiratory Tract Infection | 43
  Commonly occurring unrelated TEAE: Pyrexia: number analyzed (Participants) | 9
  Commonly occurring unrelated TEAE: Pyrexia | 16
  Commonly occurring unrelated TEAE: Cough: number analyzed (Participants) | 7
  Commonly occurring unrelated TEAE: Cough | 7
  Commonly occurring unrelated TEAE: Vomiting: number analyzed (Participants) | 6
  Commonly occurring unrelated TEAE: Vomiting | 6
  Commonly occurring unrelated TEAE: Abdominal Pain: number analyzed (Participants) | 6
  Commonly occurring unrelated TEAE: Abdominal Pain | 7
  Commonly occurring possibly related TEAE: Neutropenia/ANC Count Decreased: number analyzed (Participants) | 4
  Commonly occurring possibly related TEAE: Neutropenia/ANC Count Decreased | 4
  Commonly occurring possibly related TEAE: Thrombocytopenia/Platelet Count Decreased: number analyzed (Participants) | 3
  Commonly occurring possibly related TEAE: Thrombocytopenia/Platelet Count Decreased | 6

8. Secondary Outcome: Absolute Neutrophil Count (ANC)
Description: Safety review for haematological toxicity (mild myelosuppression target: 1-3x10^9/L)
Time Frame: Baseline and Week 60 (or final visit); max 15 months on treatment
Population: Safety population = 32 participants, who received at least one dose of oral hydroxyurea.
  Baseline value is the last non-missing assessment prior to first exposure of oral hydroxyurea.
  Week 60 is the final study visit or withdrawal at which point oral hydroxyurea was halted.
Measure: Mean (Standard Deviation); unit: x10^9 neutrophils/L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
x10^9 neutrophils/L
  Screening (Overall): number analyzed (Participants) | 31
  Screening (Overall) | 4.90 (1.825)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 5
  Screening (6 months - 1.99 years) | 4.30 (1.608)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 5.38 (2.087)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 4.43 (1.354)
  Final Visit (Overall): number analyzed (Participants) | 29
  Final Visit (Overall) | 2.70 (1.033)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 2.27 (0.671)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 2.46 (0.837)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 3.48 (1.255)

9. Secondary Outcome: White Blood Cell Count (Leukocytes)
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Baseline to Week 60 or Final Visit; max 15 months on treatment
Population: Leukocytes Safety population = 32 participants, who received at least one dose of oral hydroxyurea.
  Baseline value is the last non-missing assessment prior to first exposure of oral hydroxyurea.
  Week 60 is the final study visit or withdrawal at which point oral hydroxyurea was halted.
Measure: Mean (Standard Deviation); unit: 10^9 leukocytes/L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
10^9 leukocytes/L
  Screening (Overall): number analyzed (Participants) | 31
  Screening (Overall) | 13.01 (3.514)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 5
  Screening (6 months - 1.99 years) | 12.24 (2.019)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 14.59 (3.856)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 10.88 (2.188)
  Final Visit (Overall): number analyzed (Participants) | 29
  Final Visit (Overall) | 7.48 (2.286)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 7.90 (2.466)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 6.83 (2.244)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 8.41 (2.108)

10. Secondary Outcome: Platelets
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Baseline to Week 60 (or Final Visit), max 15 months on treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
10^9 platelets/L
  Screening (Overall): number analyzed (Participants) | 31
  Screening (Overall) | 409.06 (131.542)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 5
  Screening (6 months - 1.99 years) | 383.80 (52.756)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 381.31 (104.305)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 466.10 (181.577)
  Final Visit (Overall): number analyzed (Participants) | 29
  Final Visit (Overall) | 315.10 (134.057)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 333.67 (98.699)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 258.00 (141.782)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 408.25 (86.742)

11. Secondary Outcome: Mean Corpuscular Hemoglobin (MCH)
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Baseline to Week 60 (or Final Visit), max 15 months on treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
pg
  Screening (Overall): number analyzed (Participants) | 16
  Screening (Overall) | 27.57 (3.741)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 3
  Screening (6 months - 1.99 years) | 23.80 (3.291)
  Screening (2 - 5.99 years): number analyzed (Participants) | 7
  Screening (2 - 5.99 years) | 28.36 (4.665)
  Screening (6 - 17.99 years): number analyzed (Participants) | 6
  Screening (6 - 17.99 years) | 28.53 (1.015)
  Final Visit (Overall): number analyzed (Participants) | 27
  Final Visit (Overall) | 33.36 (4.590)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 4
  Final Visit (6 months - 1.99 years) | 28.95 (8.126)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 34.02 (3.971)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 34.31 (2.307)

12. Secondary Outcome: Hematocrit
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Up to Week 60
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: % by volume of red blood cells in blood
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
% by volume of red blood cells in blood
  Screening (Overall) | 25.02 (4.4)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 6
  Screening (6 months - 1.99 years) | 30.60 (3.161)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 23.24 (3.378)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 24.30 (4.081)
  Final Visit (Overall): number analyzed (Participants) | 27
  Final Visit (Overall) | 27.74 (3.995)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 4
  Final Visit (6 months - 1.99 years) | 30.38 (3.035)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 28.45 (4.001)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 25.10 (3.208)

13. Secondary Outcome: Bilirubin
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Up to Week 60
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
umol/L
  Screening (Overall) | 37.43 (19.649)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 6
  Screening (6 months - 1.99 years) | 14.78 (9.763)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 39.60 (19.777)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 47.53 (12.702)
  Final Visit (Overall): number analyzed (Participants) | 29
  Final Visit (Overall) | 26.12 (16.191)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 7.42 (1.941)
  Final Visit (Screening (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (Screening (2 - 5.99 years) | 26.25 (13.331)
  Final Visit (Screening (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (Screening (6 - 17.99 years) | 39.89 (13.191)

14. Secondary Outcome: Elevation in Liver Function Tests (LFTs)
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry, including Liver Function Tests (LFTs): Alkaline Phosphatase (ALP), Gamma Glutamyl Transferase (GGT), Aspartate Amino Transferase (AST), Alanine Aminotransferase (ALT)
Time Frame: Up to Week 60
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
ukat/L
  ALP Screening (Overall) | 3.55 (0.846)
  ALP Screening (6 months - 1.99 years): number analyzed (Participants) | 6
  ALP Screening (6 months - 1.99 years) | 4.19 (0.983)
  ALP Screening (2 - 5.99 years): number analyzed (Participants) | 16
  ALP Screening (2 - 5.99 years) | 3.60 (0.666)
  ALP Screening (6 - 17.99 years): number analyzed (Participants) | 10
  ALP Screening (6 - 17.99 years) | 3.10 (0.827)
  ALP Final Visit (Overall): number analyzed (Participants) | 29
  ALP Final Visit (Overall) | 3.57 (0.858)
  ALP Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  ALP Final Visit (6 months - 1.99 years) | 4.06 (0.820)
  ALP Final Visit (2 months - 5.99 years): number analyzed (Participants) | 15
  ALP Final Visit (2 months - 5.99 years) | 3.41 (0.578)
  ALP Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  ALP Final Visit (6 - 17.99 years) | 3.52 (1.237)
  GGT Screening (Overall) | 0.38 (0.333)
  GGT Screening (6 months - 1.99 years): number analyzed (Participants) | 6
  GGT Screening (6 months - 1.99 years) | 0.16 (0.034)
  GGT Screening (2 - 5.99 years): number analyzed (Participants) | 16
  GGT Screening (2 - 5.99 years) | 0.32 (0.231)
  GGT Screening (6 - 17.99 years): number analyzed (Participants) | 10
  GGT Screening (6 - 17.99 years) | 0.62 (0.437)
  GGT Final Visit (Overall): number analyzed (Participants) | 29
  GGT Final Visit (Overall) | 0.32 (0.233)
  GGT Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  GGT Final Visit (6 months - 1.99 years) | 0.16 (0.040)
  GGT Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  GGT Final Visit (2 - 5.99 years) | 0.29 (0.174)
  GGT Final Visit (6 - 17.99 years): number analyzed (Participants) | 10
  GGT Final Visit (6 - 17.99 years) | 0.49 (0.316)
  AST Screening (Overall): number analyzed (Participants) | 30
  AST Screening (Overall) | 0.85 (0.221)
  AST Screening (6 months - 1.99 years): number analyzed (Participants) | 5
  AST Screening (6 months - 1.99 years) | 0.72 (0.178)
  AST Screening (2 - 5.99 years): number analyzed (Participants) | 15
  AST Screening (2 - 5.99 years) | 0.84 (0.212)
  AST Screening (6 - 17.99 years): number analyzed (Participants) | 10
  AST Screening (6 - 17.99 years) | 0.92 (0.244)
  AST Final Visit (Overallk): number analyzed (Participants) | 29
  AST Final Visit (Overallk) | 0.67 (0.165)
  AST Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  AST Final Visit (6 months - 1.99 years) | 0.61 (0.066)
  AST Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  AST Final Visit (2 - 5.99 years) | 0.68 (0.185)
  AST Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  AST Final Visit (6 - 17.99 years) | 0.71 (0.181)
  ALT Screening (Overall) | 0.33 (0.128)
  ALT Screening (6 months - 1.99 years): number analyzed (Participants) | 6
  ALT Screening (6 months - 1.99 years) | 0.34 (0.053)
  ALT Screening (2 - 5.99 years): number analyzed (Participants) | 16
  ALT Screening (2 - 5.99 years) | 0.30 (0.129)
  ALT Screening (6 - 17.99 years): number analyzed (Participants) | 10
  ALT Screening (6 - 17.99 years) | 0.35 (0.158)
  ALT Final Visit (Overall): number analyzed (Participants) | 29
  ALT Final Visit (Overall) | 0.31 (0.110)
  ALT Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  ALT Final Visit (6 months - 1.99 years) | 0.33 (0.067)
  ALT Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  ALT Final Visit (2 - 5.99 years) | 0.30 (0.109)
  ALT Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  ALT Final Visit (6 - 17.99 years) | 0.32 (0.142)

15. Secondary Outcome: Hemoglobin
Description: Safety and efficacy of hydroxyurea therapy
Time Frame: Baseline to Week 60 (or Final Visit); max 15 months on treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
g/dL
  Screening (Overall): number analyzed (Participants) | 31
  Screening (Overall) | 8.32 (1.114)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 5
  Screening (6 months - 1.99 years) | 9.76 (0.847)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 8.07 (0.980)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 7.99 (0.911)
  Final Visit (Overall): number analyzed (Participants) | 29
  Final Visit (Overall) | 9.47 (1.369)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 10.60 (1.421)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 9.47 (1.190)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 8.63 (1.149)

16. Secondary Outcome: Bacterial Infections
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Up to Week 60
Population: Safety population = 32 participants, who received at least one dose of oral hydroxyurea.
  At screening, subjects' experiences of clinical SCA symptoms within the 12 months prior to the screening visit were recorded.
  At subsequent visits, subjects' experiences of SCA symptoms since the previous visit were recorded, until end of study.
  Each subject counted a maximum of once each per SCA symptom for before treatment and after treatment.
Measure: Number; unit: events
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
events
  Prior to Treatment (Overall) | 7
  Prior to Treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  Prior to Treatment (6 months - 1.99 years) | 0
  Prior to Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  Prior to Treatment (2 - 5.99 years) | 3
  Prior to Treatment (6 - 17.99 years): number analyzed (Participants) | 10
  Prior to Treatment (6 - 17.99 years) | 4
  After Treatment (Overall) | 17
  After Treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  After Treatment (6 months - 1.99 years) | 1
  After Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  After Treatment (2 - 5.99 years) | 8
  After Treatment (6 - 17.99 years): number analyzed (Participants) | 10
  After Treatment (6 - 17.99 years) | 8

17. Secondary Outcome: Viral Infections
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Up to Week 60
Population: At screening, subjects' experiences of clinical SCA symptoms within the 12 months prior to the screening visit were recorded.
  At subsequent visits, subjects' experiences of SCA symptoms since the previous visit were recorded, until end of study.
  Each subject counted a maximum of once each per SCA symptom for before treatment and after treatment.
Measure: Number; unit: Events
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
Events
  Prior to Treatment (Overall): number analyzed (Participants) | 26
  Prior to Treatment (Overall) | 8
  Prior to Treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  Prior to Treatment (6 months - 1.99 years) | 0
  Prior to Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  Prior to Treatment (2 - 5.99 years) | 8
  Prior to Treatment (6 - 17.99 years): number analyzed (Participants) | 10
  Prior to Treatment (6 - 17.99 years) | 0
  After Treatment (Overall) | 23
  After Treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  After Treatment (6 months - 1.99 years) | 4
  After Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  After Treatment (2 - 5.99 years) | 12
  After Treatment (6 - 17.99 years): number analyzed (Participants) | 10
  After Treatment (6 - 17.99 years) | 7

18. Secondary Outcome: Fungal Infections
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Up to Week 60
Population: as for outcome 17
Measure: Number; unit: events
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
events
  Prior to Treatment (Overall) | 1
  Prior to Treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  Prior to Treatment (6 months - 1.99 years) | 0
  Prior to Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  Prior to Treatment (2 - 5.99 years) | 0
  Prior to Treatment (6 - 17.99 years): number analyzed (Participants) | 10
  Prior to Treatment (6 - 17.99 years) | 1
  After Treatment (Overall) | 4
  After Treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  After Treatment (6 months - 1.99 years) | 1
  After Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  After Treatment (2 - 5.99 years) | 1
  After Treatment (6 - 17.99 years): number analyzed (Participants) | 10
  After Treatment (6 - 17.99 years) | 2

19. Secondary Outcome: Leg Ulcers
Description: Impact of Hydroxyurea on Safety, Hematology and Biochemistry
Time Frame: Up to Week 60
Population: as for outcome 17
Measure: Number; unit: events
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
events
  Prior to Treatment (Overall) | 0
  Prior to Treatment (6 months -1.99 years): number analyzed (Participants) | 6
  Prior to Treatment (6 months -1.99 years) | 0
  Prior to Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  Prior to Treatment (2 - 5.99 years) | 0
  Prior to Treatment (6 -17.99 years): number analyzed (Participants) | 10
  Prior to Treatment (6 -17.99 years) | 0
  After Treatment (Overall) | 1
  After Treatment (6 months -1.99 years): number analyzed (Participants) | 6
  After Treatment (6 months -1.99 years) | 0
  After Treatment (2 - 5.99 years): number analyzed (Participants) | 16
  After Treatment (2 - 5.99 years) | 0
  After Treatment (6 - 17.99 years): number analyzed (Participants) | 10
  After Treatment (6 - 17.99 years) | 1

20. Secondary Outcome: Fetal Hemoglobin
Description: Biomarker endpoints of Hydroxyurea efficacy
Time Frame: Baseline to Week 60 (or Final Visit); max 15 months on treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Hemoglobin F/Total Hemoglobin %
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
Hemoglobin F/Total Hemoglobin %
  Screening (Overall): number analyzed (Participants) | 27
  Screening (Overall) | 11.90 (8.711)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 6
  Screening (6 months - 1.99 years) | 21.52 (6.889)
  Screening (2 - 5.99 years): number analyzed (Participants) | 14
  Screening (2 - 5.99 years) | 10.94 (7.637)
  Screening (6 - 17.99 years): number analyzed (Participants) | 7
  Screening (6 - 17.99 years) | 5.57 (4.641)
  Final Visit (Overall): number analyzed (Participants) | 26
  Final Visit (Overall) | 23.53 (11.179)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 26.32 (4.893)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 14
  Final Visit (2 - 5.99 years) | 27.09 (11.888)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 6
  Final Visit (6 - 17.99 years) | 12.47 (6.467)

21. Secondary Outcome: Mean Corpuscular Volume (MCV)
Description: Biomarker endpoints of Hydroxyurea efficacy
Time Frame: Baseline to Week 60 (or Final Visit); max 15 months on treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
fL
  Screening (Overall): number analyzed (Participants) | 31
  Screening (Overall) | 83.13 (8.643)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 5
  Screening (6 months - 1.99 years) | 76.42 (7.682)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 83.25 (9.715)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 86.30 (5.410)
  Final Visit (Overall): number analyzed (Participants) | 29
  Final Visit (Overall) | 97.64 (13.700)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 81.68 (14.506)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 102.49 (11.736)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 100.51 (6.859)

22. Secondary Outcome: Cystatin C
Description: Biomarker Endpoints
Time Frame: PK1 (day 1), week 20-32 (6 months) and Week 60 (Final Visit)
Population: Baseline value is the last non-missing assessment prior to first exposure of oral HU.
  Analysis was from initiation of study drug, again at ~6months (between 20-32 weeks) and at final study visit.
  Week 28 (6 months - 1.99 years) no measures were analysed at this timepoint.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
nmol/L
  PK1 Day 1 (Overall): number analyzed (Participants) | 21
  PK1 Day 1 (Overall) | 7.52 (1.288)
  PK1 Day 1 (6 months - 1.99 years): number analyzed (Participants) | 6
  PK1 Day 1 (6 months - 1.99 years) | 8.89 (1.170)
  PK1 Day 1 (2 - 5.99 years): number analyzed (Participants) | 10
  PK1 Day 1 (2 - 5.99 years) | 6.87 (1.001)
  PK1 Day 1 (6 - 17.99 years): number analyzed (Participants) | 5
  PK1 Day 1 (6 - 17.99 years) | 7.18 (0.549)
  Week 24 (Overall): number analyzed (Participants) | 15
  Week 24 (Overall) | 7.50 (1.173)
  Week 24 (6 months - 1.99 years): number analyzed (Participants) | 4
  Week 24 (6 months - 1.99 years) | 8.36 (0.263)
  Week 24 (2 - 5.99 years): number analyzed (Participants) | 8
  Week 24 (2 - 5.99 years) | 7.07 (1.074)
  Week 24 (6 - 17.99 years): number analyzed (Participants) | 3
  Week 24 (6 - 17.99 years) | 7.52 (1.810)
  Week 28 (Overall): number analyzed (Participants) | 2
  Week 28 (Overall) | 8.67 (0.134)
  Week 28 (2 - 5.99 years): number analyzed (Participants) | 1
  Week 28 (2 - 5.99 years) | 8.76 (NA) — No SD possible when only n=1 participant analysed at this timepoint for this age group
  Week 28 (6 - 17.99 years): number analyzed (Participants) | 1
  Week 28 (6 - 17.99 years) | 8.57 (NA) — No SD possible when only n=1 participant analysed at this timepoint for this age group
  Final Visit (Overall): number analyzed (Participants) | 24
  Final Visit (Overall) | 7.44 (1.340)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 8.63 (0.999)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 11
  Final Visit (2 - 5.99 years) | 7.19 (1.253)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 7
  Final Visit (6 - 17.99 years) | 6.80 (1.192)

23. Secondary Outcome: Incidence of Acute Vaso-Occlusive Pain Crises (VOC)
Description: Hospitalization Incidence for 12 Months Prior to and After First Dose of IMP (Safety Population) for vaso-occlusive crisis (Mean [SD])
Time Frame: 12 months prior to treatment and time-averaged 12 months post-treatment; maximum 15 months on IMP
Population: Time-averaged hospitalizations after treatment was determined by dividing incidence of hospitalizations prior to treatment by 12 if study end date was more than a year after treatment start date, or by dividing by (End date - Treatment Start Date)/30.4375 otherwise. Hospitalizations did not include visits to ER/accident without hospitalization. Hospitalizations were sub-categorized by a medical monitor. Data were obtained through medical record review and study participant recall.
Measure: Mean (Standard Deviation); unit: hospitalisation events per month
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
hospitalisation events per month
  VOC 12months prior (Overall) | 0.5 (0.92)
  VOC 12months prior (6 months - 1.99 years)): number analyzed (Participants) | 6
  VOC 12months prior (6 months - 1.99 years)) | 0.0 (0.0)
  VOC 12months prior (2 - 5.99 years)): number analyzed (Participants) | 16
  VOC 12months prior (2 - 5.99 years)) | 0.7 (1.08)
  VOC 12months prior (6 - 17.99 years): number analyzed (Participants) | 10
  VOC 12months prior (6 - 17.99 years) | 0.6 (0.84)
  VOC 12months after treatment (Overall) | 0.2 (0.51)
  VOC 12months after treatment (6 months - 1.99 years)): number analyzed (Participants) | 6
  VOC 12months after treatment (6 months - 1.99 years)) | 0.3 (0.82)
  VOC 12months after treatment (2 - 5.99 years): number analyzed (Participants) | 16
  VOC 12months after treatment (2 - 5.99 years) | 0.0 (0.0)
  VOC 12months after treatment (6 - 17.99 years)): number analyzed (Participants) | 10
  VOC 12months after treatment (6 - 17.99 years)) | 0.3 (0.67)

24. Secondary Outcome: Number and Frequency of Blood Transfusions
Description: Clinical status endpoints, related to blood transfusions for treatment of SCA, this may be hospitalization, A&E, or in-clinic treatment from safety population (n=32)
Time Frame: Up to Week 60
Population: Safety population = 32 participants, who received at least one dose of oral hydroxyurea.
  Baseline value is the last non-missing assessment prior to first exposure of oral hydroxyurea.
  Week 60 is the final study visit or withdrawal at which point oral hydroxyurea was halted.
  Age group (6 months to 1.99 years) did not report any blood transfusions.
Measure: Number; unit: events (number of transfusions)
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 7
events (number of transfusions)
  Overall | 30
  2 years - 5.99 years: number analyzed (Participants) | 2
  2 years - 5.99 years | 21
  6 years - 17.99 years: number analyzed (Participants) | 5
  6 years - 17.99 years | 9

25. Secondary Outcome: Acute Chest Syndrome (ACS)
Description: Hospitalization Incidence for 12 Months Prior to and After First Dose of IMP (Safety Population) for Acute Chest Syndrome (Mean [SD])
Time Frame: 12 months prior to treatment and time averaged 12 months post-treatment; maximum 15 months on IMP
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hospitalisation events per month
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
hospitalisation events per month
  ACS Hospitalisations 12 months prior (Overall) | 0.5 (0.92)
  ACS Hospitalisations 12 months prior (6 months - 1.99 years): number analyzed (Participants) | 6
  ACS Hospitalisations 12 months prior (6 months - 1.99 years) | 0.00 (0.00)
  ACS Hospitalisations 12 months prior (2 - 5.99 years): number analyzed (Participants) | 16
  ACS Hospitalisations 12 months prior (2 - 5.99 years) | 0.6 (0.89)
  ACS Hospitalisations 12 months prior (6 - 17.99 years): number analyzed (Participants) | 10
  ACS Hospitalisations 12 months prior (6 - 17.99 years) | 0.7 (1.16)
  ACS Hospitalisations 12 months after treatment (Overall) | 0.2 (0.37)
  ACS Hospitalisations 12 months after treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  ACS Hospitalisations 12 months after treatment (6 months - 1.99 years) | 0.00 (0.00)
  ACS Hospitalisations 12 months after treatment (2 - 5.99 years): number analyzed (Participants) | 16
  ACS Hospitalisations 12 months after treatment (2 - 5.99 years) | 0.3 (0.45)
  ACS Hospitalisations 12 months after treatment (6 - 17.99 years): number analyzed (Participants) | 10
  ACS Hospitalisations 12 months after treatment (6 - 17.99 years) | 0.1 (0.32)

26. Secondary Outcome: Hospitalizations
Description: Clinical Status endpoints, all hospitalisations (not ER/Accident without hospitalization) (Mean [SD])
Time Frame: 12 months prior to treatment and time-averaged 12 months post-treatment; maximum 15 months on IMP
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hospitalisation events per month
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
hospitalisation events per month
  Hospitalisations 12 months prior (Overall) | 1.7 (1.54)
  Hospitalisations 12 months prior (6 months - 1.99 years): number analyzed (Participants) | 6
  Hospitalisations 12 months prior (6 months - 1.99 years) | 0.3 (0.82)
  Hospitalisations 12 months prior (2 - 5.99 years): number analyzed (Participants) | 16
  Hospitalisations 12 months prior (2 - 5.99 years) | 2.0 (1.59)
  Hospitalisations 12 months prior (6 - 17.99 years): number analyzed (Participants) | 10
  Hospitalisations 12 months prior (6 - 17.99 years) | 1.9 (1.45)
  Hospitalisations 12 months after treatment (Overall) | 0.3 (0.65)
  Hospitalisations 12 months after treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  Hospitalisations 12 months after treatment (6 months - 1.99 years) | 0.3 (0.82)
  Hospitalisations 12 months after treatment (2 - 5.99 years): number analyzed (Participants) | 16
  Hospitalisations 12 months after treatment (2 - 5.99 years) | 0.3 (0.45)
  Hospitalisations 12 months after treatment (6 - 17.99 years): number analyzed (Participants) | 10
  Hospitalisations 12 months after treatment (6 - 17.99 years) | 0.5 (0.85)

27. Secondary Outcome: Dose Escalation i.e. Maximum Tolerated Dose (MTD)
Description: Summary of maximum tolerated dose achieved in mg/kg (Mean [SD])
Time Frame: Screening Up to Final Visit (Week 60 or Withdrawal), maximum 15 months on IMP
Population: Clinical status endpoints; Safety population = 32 participants, who received at least one dose of IMP.
  Week 60 is the final study visit, or withdrawal point at which point IMP was halted.
  MTD only summarized for subjects who investigator denoted as achieving MTD during the study (n=20). If several doses were marked as MTD for the subject, the highest dose was used.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
mg/kg
  MTD (Overall) | 25.63 (6.780)
  MTD (6 months - 1.99 years): number analyzed (Participants) | 5
  MTD (6 months - 1.99 years) | 23.50 (8.944)
  MTD (2 - 5.99 years): number analyzed (Participants) | 9
  MTD (2 - 5.99 years) | 26.11 (5.465)
  MTD (6 - 17.99 years): number analyzed (Participants) | 6
  MTD (6 - 17.99 years) | 26.67 (7.528)

28. Secondary Outcome: Other SCA-related Hospitalizations
Description: Clinical parameters (symptoms), secondary clinical status endpoints (not including ACS, VOC, Other Non-SCA related) (mean [SD])
Time Frame: 12 months prior to treatment and time averaged 12 months post-treatment; maximum 15 months on IMP
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hospitalisation events per month
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
hospitalisation events per month
  Other SCA related Hospitalizations 12 months prior (Overall) | 0.4 (0.67)
  Other SCA related Hospitalizations 12 months prior (6 months - 1.99 years): number analyzed (Participants) | 6
  Other SCA related Hospitalizations 12 months prior (6 months - 1.99 years) | 0.3 (0.82)
  Other SCA related Hospitalizations 12 months prior (2 - 5.99 years): number analyzed (Participants) | 16
  Other SCA related Hospitalizations 12 months prior (2 - 5.99 years) | 0.4 (0.63)
  Other SCA related Hospitalizations 12 months prior (6 - 17.99 years): number analyzed (Participants) | 10
  Other SCA related Hospitalizations 12 months prior (6 - 17.99 years) | 0.4 (0.70)
  Other SCA related Hospitalizations 12 months after treatment (Overall) | 0.0 (0.18)
  Other SCA related Hospitalizations 12 months after treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  Other SCA related Hospitalizations 12 months after treatment (6 months - 1.99 years) | 0.00 (0.00)
  Other SCA related Hospitalizations 12 months after treatment (2 - 5.99 years): number analyzed (Participants) | 16
  Other SCA related Hospitalizations 12 months after treatment (2 - 5.99 years) | 0.00 (0.00)
  Other SCA related Hospitalizations 12 months after treatment (6 - 17.99 years): number analyzed (Participants) | 10
  Other SCA related Hospitalizations 12 months after treatment (6 - 17.99 years) | 0.1 (0.32)

29. Secondary Outcome: Parent/Caregiver Palatability and Acceptability Questionnaire
Description: Clinical status endpoints. Visual Analogue scale used to determine, taste, smell, aftertaste, acceptability and ease of dosing (1-100mm scale) with 1 being worst possible and 100 being best possible.
  Assessed for <6 years of age by parents/guardians. Assessed for >6 years of age, combination of parent/guardian and participant responses.
Time Frame: Taken once at any point after 8 weeks on study medication (or at early Withdrawal)
Population: Results are presented for all 32 safety participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
mm
  Taste (Overall) | 84.2 (26.21)
  Taste (6 months - 1.99 years): number analyzed (Participants) | 6
  Taste (6 months - 1.99 years) | 71.3 (23.30)
  Taste (2 - 5.99 years): number analyzed (Participants) | 16
  Taste (2 - 5.99 years) | 91.1 (23.86)
  Taste (6 - 17.99 years): number analyzed (Participants) | 10
  Taste (6 - 17.99 years) | 80.8 (30.14)
  Smell (Overall) | 83.8 (21.73)
  Smell (6 months - 1.99 years): number analyzed (Participants) | 6
  Smell (6 months - 1.99 years) | 74.8 (25.51)
  Smell (2 - 5.99 years): number analyzed (Participants) | 16
  Smell (2 - 5.99 years) | 87.5 (17.26)
  Smell (6 - 17.99 years): number analyzed (Participants) | 10
  Smell (6 - 17.99 years) | 83.1 (26.28)
  Aftertaste (>6 years): number analyzed (Participants) | 5
  Aftertaste (>6 years) | 67.6 (23.21)

30. Secondary Outcome: Vitamin D
Description: Biochemistry
Time Frame: From Screening Up to Final Visit (Week 60 or WD)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
nmol/L
  Screening (Overall) | 59.35 (32.613)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 6
  Screening (6 months - 1.99 years) | 83.07 (32.329)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 65.43 (29.076)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 35.39 (24.403)
  Final Visit (Overall): number analyzed (Participants) | 29
  Final Visit (Overall) | 62.26 (30.220)
  Final Visit (6 months - 1.99 years): number analyzed (Participants) | 6
  Final Visit (6 months - 1.99 years) | 86.44 (25.475)
  Final Visit (2 - 5.99 years): number analyzed (Participants) | 15
  Final Visit (2 - 5.99 years) | 57.54 (34.093)
  Final Visit (6 - 17.99 years): number analyzed (Participants) | 8
  Final Visit (6 - 17.99 years) | 52.97 (14.749)

31. Secondary Outcome: Other Non-SCA-related Hospitalizations
Description: Clinical parameters (symptoms), secondary clinical status endpoints (not including ACS, VOC, Other SCA-related)
Time Frame: 12 months prior to treatment and 12 months post-treatment; maximum 15 months on IMP
Population: Hospitalizations 'Prior to Treatment' having a start date within 1 year prior to initial treatment. Hospitalizations 'After Treatment' defined as all hospitalizations (not ER/Accident without hospitalization) within 1 year after treatment start date.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
events
  Other Non-SCA related Hospitalizations 12 months prior (Overall) | 0.2 (0.47)
  Other Non-SCA related Hospitalizations 12 months prior (6 months - 1.99 years): number analyzed (Participants) | 6
  Other Non-SCA related Hospitalizations 12 months prior (6 months - 1.99 years) | 0.00 (0.00)
  Other Non-SCA related Hospitalizations 12 months prior (2 - 5.99 years): number analyzed (Participants) | 16
  Other Non-SCA related Hospitalizations 12 months prior (2 - 5.99 years) | 0.3 (0.58)
  Other Non-SCA related Hospitalizations 12 months prior (6 - 17.99 years): number analyzed (Participants) | 10
  Other Non-SCA related Hospitalizations 12 months prior (6 - 17.99 years) | 0.2 (0.42)
  Other Non-SCA related Hospitalizations 12 months after treatment (Overall) | 0.00 (0.00)
  Other Non-SCA related Hospitalizations 12 months after treatment (6 months - 1.99 years): number analyzed (Participants) | 6
  Other Non-SCA related Hospitalizations 12 months after treatment (6 months - 1.99 years) | 0.00 (0.00)
  Other Non-SCA related Hospitalizations 12 months after treatment (2 - 5.99 years): number analyzed (Participants) | 16
  Other Non-SCA related Hospitalizations 12 months after treatment (2 - 5.99 years) | 0.00 (0.00)
  Other Non-SCA related Hospitalizations 12 months after treatment (6 - 17.99 years): number analyzed (Participants) | 10
  Other Non-SCA related Hospitalizations 12 months after treatment (6 - 17.99 years) | 0.00 (0.00)

32. Other Pre Specified Outcome: Transcranial Doppler Velocity
Description: Exploratory Endpoint; clinical output of hydroxyurea treatment
Time Frame: Baseline to Week 40-56 (Follow up scan).
Population: Time Averaged Mean Maximum Velocity (TAMV) in cm/sec at Baseline and Week 40-56 Visit (Safety Population).
  max 15 months on treatment at Week 60.
  Only participants with non-missing values at screening and end of study are included in the Baseline shift summary (change from baseline).
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Oral Hydroxyurea
Number analyzed (Participants) | 32
cm/sec
  Screening (Overall): number analyzed (Participants) | 30
  Screening (Overall) | 141.5 (34.71)
  Screening (6 months - 1.99 years): number analyzed (Participants) | 4
  Screening (6 months - 1.99 years) | 90.5 (9.33)
  Screening (2 - 5.99 years): number analyzed (Participants) | 16
  Screening (2 - 5.99 years) | 150.0 (34.78)
  Screening (6 - 17.99 years): number analyzed (Participants) | 10
  Screening (6 - 17.99 years) | 148.3 (22.42)
  Week 40-56 (Overall): number analyzed (Participants) | 23
  Week 40-56 (Overall) | 133.7 (26.52)
  Week 40-56 (6 months - 1.99 years): number analyzed (Participants) | 3
  Week 40-56 (6 months - 1.99 years) | 95.7 (15.18)
  Week 40-56 (2 - 5.99 years): number analyzed (Participants) | 13
  Week 40-56 (2 - 5.99 years) | 138.6 (24.86)
  Week 40-56 (6 - 17.99 years): number analyzed (Participants) | 7
  Week 40-56 (6 - 17.99 years) | 140.7 (20.79)
  Baseline Shift (Overall): number analyzed (Participants) | 21
  Baseline Shift (Overall) | -11.5 (20.74)
  Baseline Shift (6 months - 1.99 years): number analyzed (Participants) | 1
  Baseline Shift (6 months - 1.99 years) | -1.0 (NA) — Insufficient sample size.
  Baseline Shift (2 - 5.99 years): number analyzed (Participants) | 13
  Baseline Shift (2 - 5.99 years) | -13.7 (22.02)
  Baseline Shift (6 - 17.99 years): number analyzed (Participants) | 7
  Baseline Shift (6 - 17.99 years) | -9.0 (20.68)

ADVERSE EVENTS:
Time Frame: Screening to safety follow up call at 64 weeks (maximum 15 months on treatment).
Description: Protocol definition of SAE for SCA associated complications, AEs only became reportable SAEs if the hospital admission was prolonged >7days. SCA related hospitalisations <7days recorded as AEs due to the frequency of admissions within population and chronic nature of the condition. Attendance of emergency room without admission or for elective procedures were not considered SAEs unless prolonged. All SAEs unrelated to SCA condition were reportable in line with standard definitions.
Arm/Group | Oral Hydroxyurea
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 6/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Hydroxyurea (N=32)
Acute Chest Syndrome (ACS) Grade 3 (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Grade 3, requiring hospitalisation >7days (n=3 participants)
Acute Chest Syndrome (ACS) Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 2, requiring hospitalisation >7days
Vaso-occlusive Crisis (VOC) (Blood and lymphatic system disorders) | 2 (2) — Grade 3, requiring hospitalisation >7days (n=2 participants)
Anemia secondary to SCD (Blood and lymphatic system disorders) | 1 (1) — Grade 3, requiring hospitalisation for oxygen therapy and blood transfusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Hydroxyurea (N=32)
Anemia (Blood and lymphatic system disorders) | 1 (1) — *Related Treatment Emergent Adverse Event (TEAE) in Safety population (n=32). Where relatedness is defined as anything at least possibly related to the IMP.
Neutropenia/Low ANC Count (Blood and lymphatic system disorders) | 4 (4) — Haematological toxicity (ANC <1.0x10^9/L). n=3 Grade 3 events in n=3 participants; n=4 events in n=4 participants at least possibly related. In n=3 in the 6month-1.99 year age group, associated with viral/other illness or dose titration.
Thrombocytopenia/Low Platelet Count (Blood and lymphatic system disorders) | 5 (7) — Haematological toxicity (Platelet <80x10^9/L) were </= Grade 2. Of which n=6 events were considered possibly related (in 3 participants), with n=5 events in the 6 month-1.99 year age group, associated with viral/other illness or dose titration.
Haemoglobin (Hb) Decreased (Investigations) | 2 (3) — Haematological toxicity (Hb <4.5g/dL or 20% drop). n=1 event Grade 3 in n=1 participant; n=2 events at least possibly related in n=1 participant in the 6month-1.99 year age group.
Absolute Reticulocyte Count (ARC) Decreased (Investigations) | 1 (2) — Haematological toxicity (ARC <80x10^9/L; unless Hb >9.0g/dL). All events </= Grade 2; n=2 events at least possibly related in n=1 participant in the 6month-1.99 year age group.
Red Blood Cell (RBC) Count Decreased (Investigations) | 1 (2) — *Related Treatment Emergent Adverse Event (TEAE) in Safety population (n=32). Where relatedness is defined as anything at least possibly related to the IMP.
Gamma-Glutamyltransferase (GGT) Increased (Investigations) | 1 (1) — *Related Treatment Emergent Adverse Event (TEAE) in Safety population (n=32). Where relatedness is defined as anything at least possibly related to the IMP.
Hematocrit (HCT) Decreased (Investigations) | 1 (2) — *Related Treatment Emergent Adverse Event (TEAE) in Safety population (n=32). Where relatedness is defined as anything at least possibly related to the IMP.
Diarrhoea (Gastrointestinal disorders) | 4 (5) — Diarrhoea; n=1 event at least possibly related in n=1 participant; n=4 unrelated event of mild/moderate severity in n=3 participants.
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — *Related Treatment Emergent Adverse Event (TEAE) in Safety population (n=32). Where relatedness is defined as anything at least possibly related to the IMP.
Nail Discolouration (Skin and subcutaneous tissue disorders) | 1 (1) — *Related Treatment Emergent Adverse Event (TEAE) in Safety population (n=32). Where relatedness is defined as anything at least possibly related to the IMP.
Rash (Skin and subcutaneous tissue disorders) | 3 (3) — Rash; n=1 at least possibly related event in n= 1 participant; n=2 unrelated events in n=2 participants of mild/moderate severity.
Rash Papular (Skin and subcutaneous tissue disorders) | 2 (2) — *Related Treatment Emergent Adverse Event (TEAE) in Safety population (n=32). Where relatedness is defined as anything at least possibly related to the IMP.
Sickle Cell Anemia with Crisis/Vaso-Occlusive Crisis (VOC) (Blood and lymphatic system disorders) | 18 (53) — 'SCA with crisis' interchangeable with 'Vaso-Occlusive crisis (VOC).' n=7 events were Grade 3 or above in n=4 participants and did not meet the protocol definition of SAEs; Remainder n=46 in n=14 participants were mild/moderate severity.
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) — Unrelated viral URTI; n=1 Grade 3 event in 1 participant (6months -2.99years); n=2 events in n=2 participants of mild/moderate severity.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) — Unrelated pain in extremity; n=1 event Grade 3 in n=1 participant; n=4 events Grade </=2 in 4 participants.
Acute Chest Syndrome (ACS) (Respiratory, thoracic and mediastinal disorders) | 2 (3) — ACS events of mild/moderate severity unrelated to IMP that did not meet the protocol definition of SAE.
Hypereosinophilic Syndrome (Blood and lymphatic system disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Ear Pain (Ear and labyrinth disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Abdominal Pain (Gastrointestinal disorders) | 6 (7) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Constipation (Gastrointestinal disorders) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Gastritis (Gastrointestinal disorders) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Salivary Gland Enlargement (Gastrointestinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Teething (Gastrointestinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Vomiting (Gastrointestinal disorders) | 6 (6) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Feeling Abnormal (General disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Influenza Like Illness (General disorders) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Injection Site Pain (General disorders) | 1 (4) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Injection Site Swelling (General disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Peripheral Swelling (General disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Pyrexia (General disorders) | 9 (16) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Swelling Face (General disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Ulcer (General disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Cholecystitis (Hepatobiliary disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Hepatomegaly (Hepatobiliary disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Drug Hypersensitivity (Immune system disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Body Tinea (Infections and infestations) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Chronic Sinusitis (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Conjunctivitis (Infections and infestations) | 3 (3) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Conjunctivitis Viral (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
COVID-19 (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Croup Infectious (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Ear Infection (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Fungal Skin Infection (Infections and infestations) | 1 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Gastroenteritis (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Gingival Abscess (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Gingivitis (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Hand-Foot-And-Mouth Disease (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Localised Infection (Infections and infestations) | 1 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Lower Respiratory Tract Infection (Infections and infestations) | 5 (5) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Nasopharyngitis (Infections and infestations) | 3 (4) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Otitis Media (Infections and infestations) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Pharyngitis (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Pharyngotonsillitis (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Rhinitis (Infections and infestations) | 3 (4) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Sinusitis (Infections and infestations) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Tinea Capitis (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Tonsilitis (Infections and infestations) | 3 (3) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Upper Respiratory Tract Infection (Infections and infestations) | 17 (43) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Urinary Tract Infection (Infections and infestations) | 2 (3) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Viral Infection (Infections and infestations) | 5 (7) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Viral Pharyngitis (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Viral Rash (Infections and infestations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Contusion (Injury, poisoning and procedural complications) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Lip Injury (Injury, poisoning and procedural complications) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Skin Laceration (Injury, poisoning and procedural complications) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Soft Tissue Injury (Injury, poisoning and procedural complications) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Alanine Aminotransferase Increased (Investigations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Aspartate Aminotransferase Increased (Investigations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Blood Iron Decreased (Investigations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Body Temperature Increased (Investigations) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Platelet Count Increased (Investigations) | 1 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Vitamin D Decreased (Investigations) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Soft Tissue Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Benign Rolandic Epilepsy (Nervous system disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Headache (Nervous system disorders) | 4 (8) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Lethargy (Nervous system disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Pica (Psychiatric disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Balanoposthitis (Reproductive system and breast disorders) | 1 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Priapism (Reproductive system and breast disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Allergic Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (7) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (3) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (4) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Skin Erosion (Skin and subcutaneous tissue disorders) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Urticaria Papular (Skin and subcutaneous tissue disorders) | 2 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Tooth Extraction (Surgical and medical procedures) | 1 (1) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.
Toothache (Gastrointestinal disorders) | 1 (2) — Unrelated Treatment Emergent (TEAEs) of mild/moderate severity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or sub-set analysis of data based on the results obtained shall not be made before the first publication by the Sponsor, in which the Investigators may be named as authors. After initial publication material for public dissemination will be submitted to the Sponsor for review at least 60 days prior to submission, where all reasonable comments by the Sponsor will be incorporated. Sponsor may request additional delay for up to 6 months to protect proprietary information/IP.

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT03763656/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT03763656/SAP_001.pdf